CLINICAL TRIAL: NCT01952938
Title: Outcome EnduRo Versus LINK SL Rotating Hinge Knee
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Orthopaedische Klinik Koenig-Ludwig-Haus (Other)
Responsible Party: Sponsor
Other Study IDs: AAG-I-H-1112
Record Dates: First submitted 2013-09-25; First posted 2013-09-30 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Knee Arthrosis,
Keywords: knee revision surgery,; rotating hinge prosthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- LINK SL: Patients
  Interventions: Procedure: LINK SL versus EnduRo
- EnduRo: Patients
  Interventions: Procedure: LINK SL versus EnduRo

INTERVENTIONS:
Procedure: LINK SL versus EnduRo

SUMMARY:
Randomized clinical outcome study of two rotating hinge knee prosthesis in knee surgery. Hypothesis: No difference in the clinical outcome for 1 year after the operation. Clinical follow-ups at 3, 10, 90 and 360 days after surgery. Measurement of clinical parameters

ELIGIBILITY:
Inclusion Criteria:

* rotating hinge knee indicated

Exclusion Criteria:

* infection,
* malignant tumor,
* rheumatism

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients need hinged knee prosthesis
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Oxford knee score | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopeadische Klinik KLH, Würzburg, Bavaria, Germany